CLINICAL TRIAL: NCT01987648
Title: E-CRANIO Trial Study on Elective CRAniotomies: Postoperative Neurointensive Care, Imaging and Outcome
Brief Title: eCRANIO Trial Study on Elective CRAniotomies: Postoperative Neurointensive Care, Imaging and Outcome
Acronym: eCRANIO
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 13-058
Record Dates: First submitted 2013-11-12; First posted 2013-11-19 (Estimated); Last update posted 2021-12-08 (Actual); Status verified 2021-12

CONDITIONS: Craniotomy; Postoperative Complications
Keywords: Craniotomy; Postoperative complications; Perioperative care; Postoperative intracerebral hemorrhage; Postoperative seizure
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All study participants: Included are all patients who 18 years or older, who get an elective craniotomy (no biopsy, no awake surgery, no re-operation) and who are treated at the Department of Neurosurgery
  Interventions: Procedure: Elective Craniotomy Patients

INTERVENTIONS:
Procedure: Elective Craniotomy Patients — Patients who receive an elective craniotomy (no biopsy, no awake surgery, no re-operation)

SUMMARY:
Regarding the postoperative care strategies following elective craniotomy procedures there is little evidence. Many neurosurgical departments prefer these patients to remain intubated and sedated for many hours postoperatively to minimize hemodynamic and respiratory distress in fear of early postoperative complications such as rebleeding or seizures. In this prospective observational study the investigators aim to show that early tracheal extubation following elective brain surgery is feasible and safe.

DETAILED DESCRIPTION:
Background

Amongst many surgical subspecialties particularly the field of neurosurgery has made major advancements in the last decade in regards to microsurgical techniques such as continuously pushing the boundaries of radical tumor resection while ensuring patient security and functional integrity nonetheless to mention just one aspect. However, once the surgeon has closed up and the patient is transferred to the intensive care or intermediate care unit for observation for the crucial early postoperative hours the brain tissue is exposed to hemodynamic and respirational changes.

Early postoperative bleeding and brain swelling are the most feared complications after elective craniotomy in neurosurgery. Unfortunately, there is no bedside monitoring to diagnose these complications at a very early state. Patients become symptomatic by a clinical neurological deterioration or an early postoperative seizure. Therefore, much attention has been paid to provide a close monitoring and observation of the patient usually at a critical care unit during the first hours after brain surgery.

Although not substantiated by hard evidence, the major postoperative strategies are the following:

1. Parameter oriented: Periods of arterial hypertension, hypoventilation with arterial CO2 increase, low oxygen saturation, extensive coughing, pressing, and pain are strictly avoided. In order to achieve this goal the patient remains intubated and sedated during the first hours postoperatively.
2. Symptom oriented: The awakened patient is monitored clinically as early as possible for a deterioration of consciousness, seizure or the development of a new neurological deficit. Thus, the patient is extubated in a timely fashion postoperatively.

Evidently, both strategies are opposite to each other, since strategy 1 requires keeping the patient sedated and intubated over a longer period of time and weaning from artificial ventilation is performed at the critical care unit. This hinders early diagnosis of a neurological deterioration and timely action. On the contrary, strategy 2 aims at a very early extubation of the patient immediately after completing the surgical procedure, which exposes the patient to more hemodynamic and cardiopulmonary stress which may lead to a higher likelihood of a secondary neurological injury.

Since, to the best of the investigators' knowledge, there is no prospective data, depending on the philosophy of the neurosurgeon, the anesthetist and the neuro-intensivist one strategy is preferred over another. For this clinical study, the Department of Neurosurgery Berne is conducting a prospective observational study to show that early tracheal extubation following elective brain surgery is feasible and safe.

Objective

The investigators aim to provide prospective data with respect to complications of early extubation and to compare these results to existing data in the literature with the delayed extubation strategy after elective craniotomy. The investigators believe early extubation and continuous clinical monitoring does not coincide with a higher rate of postoperative complications. Furthermore, strategy 2 might even be superior to strategy 1 in that respect. Also, by conducting this clinical trial the investigators hope to get a more profound insight to further improve the postoperative patient management after elective brain surgery.

The primary endpoint is the incidence of significant postoperative intracranial hemorrhage, brain swelling or seizure leading to either surgical intervention or any new, secondary neurological deficit, coma, palliative care or death related to postoperative events.

As a secondary endpoint the investigators will assess the role of routine early postoperative CT imaging before transfer to the ward and surgical drains.

Methods

This clinical study is designed as a prospective monocenter observational trial. Data as defined in a case report form will be collected of patients undergoing elective craniotomy at the departments of neurosurgery of the University Hospitals in Bern. Patient data collection begins at admission and ends at hospital discharge except for a mortality follow-up of 30 days postoperatively. Statistical analysis will be performed as defined in the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* 18 Years and older
* Elective craniotomy for any mass lesion or vascular lesion
* Early extubation

Exclusion Criteria

* Biopsy only
* Re-operation
* Craniotomy due to infection
* Awake surgery/craniotomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who 18 years or older,who get an elective craniotomy (no biopsy, no awake surgery, no re-operation) and who are treated at the Department of Neurosurgery
Sampling Method: Probability Sample
Enrollment: 1969 (Actual)
Dates: Start 2011-11-01 (Actual); Primary Completion 2021-09-28 (Actual); Study Completion 2021-10 (Actual)

PRIMARY OUTCOMES:
Morbidity | 48 hours postoperative

SECONDARY OUTCOMES:
Re-Intubation | 48 hours postoperative
Mortality | 30 Days
Emergency CT Scan | 48 hours postoperative
Re Operation | 48 hours postoperative
Length of postoperative stay on ICU and IMC | 30 Days

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Schär, MD, Principal Investigator — Department of Neurosurgery, Inselspital Berne; Jürgen Beck, Prof., Study Chair — Department of Neurosurgery, Inselspital Berne
Locations (1):
- University Berne, Department of Neurosurgery, Bern, Switzerland

REFERENCES:
- [Background] Basali A, Mascha EJ, Kalfas I, Schubert A. Relation between perioperative hypertension and intracranial hemorrhage after craniotomy. Anesthesiology. 2000 Jul;93(1):48-54. doi: 10.1097/00000542-200007000-00012. PMID 10861145
- [Background] Fadul C, Wood J, Thaler H, Galicich J, Patterson RH Jr, Posner JB. Morbidity and mortality of craniotomy for excision of supratentorial gliomas. Neurology. 1988 Sep;38(9):1374-9. doi: 10.1212/wnl.38.9.1374. PMID 3412585
- [Background] Flint AC, Manley GT, Gean AD, Hemphill JC 3rd, Rosenthal G. Post-operative expansion of hemorrhagic contusions after unilateral decompressive hemicraniectomy in severe traumatic brain injury. J Neurotrauma. 2008 May;25(5):503-12. doi: 10.1089/neu.2007.0442. PMID 18346002
- [Background] Fukamachi A, Koizumi H, Nagaseki Y, Nukui H. Postoperative extradural hematomas: computed tomographic survey of 1105 intracranial operations. Neurosurgery. 1986 Oct;19(4):589-93. doi: 10.1227/00006123-198610000-00013. PMID 3785596
- [Background] Fukamachi A, Koizumi H, Nukui H. Postoperative intracerebral hemorrhages: a survey of computed tomographic findings after 1074 intracranial operations. Surg Neurol. 1985 Jun;23(6):575-80. doi: 10.1016/0090-3019(85)90006-0. PMID 3992457
- [Background] Gerald AG. Update on hemostasis: neurosurgery. Surgery. 2007 Oct;142(4 Suppl):S55-60. doi: 10.1016/j.surg.2007.06.030. PMID 18019938
- [Background] Kalfas IH, Little JR. Postoperative hemorrhage: a survey of 4992 intracranial procedures. Neurosurgery. 1988 Sep;23(3):343-7. doi: 10.1227/00006123-198809000-00010. PMID 3226512
- [Background] Merriman E, Bell W, Long DM. Surgical postoperative bleeding associated with aspirin ingestion. Report of two cases. J Neurosurg. 1979 May;50(5):682-4. doi: 10.3171/jns.1979.50.5.0682. PMID 430164
- [Background] Morgan MK, Johnston IH, Hallinan JM, Weber NC. Complications of surgery for arteriovenous malformations of the brain. J Neurosurg. 1993 Feb;78(2):176-82. doi: 10.3171/jns.1993.78.2.0176. PMID 8421199
- [Background] Palmer JD, Sparrow OC, Iannotti F. Postoperative hematoma: a 5-year survey and identification of avoidable risk factors. Neurosurgery. 1994 Dec;35(6):1061-4; discussion 1064-5. doi: 10.1227/00006123-199412000-00007. PMID 7885549
- [Derived] Schar RT, Tashi S, Branca M, Soll N, Cipriani D, Schwarz C, Pollo C, Schucht P, Ulrich CT, Beck J, Z'Graggen WJ, Raabe A. How safe are elective craniotomies in elderly patients in neurosurgery today? A prospective cohort study of 1452 consecutive cases. J Neurosurg. 2020 Apr 24;134(3):1113-1121. doi: 10.3171/2020.2.JNS193460. Print 2021 Mar 1. PMID 32330879
- [Derived] Schar RT, Fiechter M, Z'Graggen WJ, Soll N, Krejci V, Wiest R, Raabe A, Beck J. No Routine Postoperative Head CT following Elective Craniotomy--A Paradigm Shift? PLoS One. 2016 Apr 14;11(4):e0153499. doi: 10.1371/journal.pone.0153499. eCollection 2016. PMID 27077906